CLINICAL TRIAL: NCT03340610
Title: Intravitreal Alflibercept Injection (IAI) for Persistent Diabetic Macular Edema (DME) After Treatment With Bevacizumab And Ranibizumab
Brief Title: IAI for Persistent DME After Treatment With Bevacizumab And Ranibizumab
Acronym: ROTATED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Southeast Retina Center, Georgia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFTe-DME-1519
Record Dates: First submitted 2017-11-08; First posted 2017-11-13 (Actual); Results first posted 2019-05-01 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open Label Single Arm Trial (Other): Evaluating the efficacy of Alflibercept Injections in DME Following Treatment With Bevacizumab and Ranibizumab
  Interventions: Drug: Alflibercept

INTERVENTIONS:
Drug: Alflibercept — Intravitreal Injection
  Other Names: Eylea

SUMMARY:
This is a phase 4 prospective, nonrandomized, open label, interventional clinical trial. Study eyes will receive 5 required initial monthly Intravitreal Aflibercept (IAI) doses of 2 mg followed by 2q8 IAI for a total of 52 weeks; only one study eye from each patient will be enrolled.

DETAILED DESCRIPTION:
This is a phase 4 prospective, nonrandomized, open label, interventional clinical trial. Study eyes will receive 5 required initial monthly IAI doses of 2 mg followed by 2q8 IAI for a total of 52 weeks; only one study eye from each patient will be enrolled.

Starting at week 24, patients may be eligible to receive additional 2mg IAI (2q4) treatment if both of the following criteria is met and the investigator feels additional treatment would be beneficial:

* Loss of >5 letters from baseline or best previously recorded best corrected visual acuity (BCVA)
* Presence of new or recurrent intraretinal fluid or subretinal fluid as assessed by SD OCT

Starting at week 24, rescue therapy with macular laser photocoagulation may be administered if any the following criteria are met

* Loss of > 15 letters from baseline or best previously recorded BCVA and loss of acuity felt to be secondary to Diabetic Macular Edema (DME) and not from other cause (i.e., cataract, epiretinal membrane, vitreous hemorrhage, etc) and investigator feels patient would benefit from rescue therapy
* Increase in SD OCT CSF > 100 um from baseline or best previously recorded SD OCT CSF and investigator feels patient would benefit from rescue therapy.

Every 4 week visit will include ETDRS BCVA, IOP measurement, Slit lamp biomicroscopy, Indirect ophthalmoscopy, Heidelberg Spectralis SD-OCT and evaluation for systemic and ocular adverse events. Fundus Photography and Wide field Optos fluorescein angiography will be performed at baseline and at week 20and week 52.

STUDY DURATION: Approximately 52 weeks to the end of the study. Primary endpoint will be evaluated at week 52.

ELIGIBILITY:
Inclusion Criteria:

A patient must meet the following criteria to be eligible for inclusion in the study:

1. Adults with Diabetes Mellitus 2. Documented history of ROTATE study completion (within 3 months +/- 1 week of exit visit) 3. BCVA ETDRS visual acuity letter score 20/25-20/400 4. Thickening due to DME involving the center of the macula evident on clinical exam 5. DME on OCT at baseline (>305 microns if male or >290 microns if female) as assessed on Heidelberg Spectralis SD OCT 6. At least 30 days but less than 45 days since prior 0.3 mg ranibizumab injection 7. Willing and able to comply with clinic visits and study-related procedures 8. Provide signed HIPAA statement and informed consent prior to any study procedures

-

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from the study:

1. Macular edema considered to be due to a cause other than DME (ERM, Vein Occlusion, Postop CME, uveitis)
2. History of PRP within 3 months prior to enrollment or anticipated need for PRP
3. History of idiopathic or autoimmune uveitis in the study eye
4. Cataract surgery in the study eye within 90 days of baseline
5. Any intraocular surgery within 90 days of baseline
6. Vitreomacular traction or epiretinal membrane in the study eye that is thought to affect vision
7. Clinically significant pre-retinal fibrosis involving the macula in the study eye per investigator judgment
8. Intraocular inflammation of trace or above in the study eye
9. Evidence of active infection in either eye
10. Uncontrolled glaucoma in the study eye defined as a pressure of > 25 on maximal medical therapy.
11. Concurrent disease in the study eye, other than DME, that could compromise VA, require medical or surgical intervention during the study or could confound interpretation of the results
12. Ocular media of insufficient quality to obtain fundus and OCT images
13. Current treatment for a serious systemic infection
14. Administration of systemic anti-angiogenic agents within 180 days of screen
15. History of yag capsulotomy within 1 month prior to enrollment
16. Receipt of any treatment for DME, other than ranibizumab 0.3 mg, in the study eye at any time in the past 3 months following ROTATE study exit, (such as focal/grid macular photocoagulation, intravitreal or peribulbar corticosteroids or other anti-VEGF agents such as Macugen, 2 mg IAI,, 0.5 mg ranibizumab, or intravitreal bevacizumab)
17. Any women who are pregnant, breast-feeding, or attempting to become pregnant
18. Sexually active men* or women of childbearing potential** who are unwilling to practice adequate contraception during the study (adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device [IUD]; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly)

    * Contraception is not required for men with documented vasectomy. **Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of child bearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis M Marcus, MD, Principal Investigator — Southeast Retina Center, PC.
Locations (1):
- Southeast Retina Center, Augusta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 4 Prospective, Nonrandomized, Open Label, Interventional: Evaluating the efficacy of Alflibercept Injections in DME Following Treatment With Bevacizumab and Ranibizumab
  Alflibercept: Intravitreal Injection
  Study eyes will receive 5 required initial monthly IAI doses of 2 mg followed by 2q8 IAI for a total of 52 weeks.
Period: Overall Study
Arm/Group | Phase 4 Prospective, Nonrandomized, Open Label, Interventional
Started | 30
Completed | 27
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Single Arm Trial
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 15
Age, Continuous [Mean (Full Range); unit: years] | 63 [43 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
Insulin Dependency (Independent/Dependent) [Count of Participants; unit: Participants]
  Independent | 13
  Dependent | 17
Diabetic Retinopathy (Proliferative/Non-Proliferative) [Count of Participants; unit: Participants]
  Proliferative | 11
  Non-Proliferative | 19
Average Anti-VEGF Injections Received Prior to Baseline [Mean (Full Range); unit: injections] | 14.5 [6 to 48]
Baseline Visual Acuity [Mean (Full Range); unit: letters] | 64 [36 to 83]
Baseline Optical Coherence Tomography (OCT) Central Subfield Thickness (CST) [Mean (Full Range); unit: microns] | 459 [310 to 721]
Eyes with Prior Macular Laser [Count of Participants; unit: Participants] | 7
Eyes with Prior Panretinal Photocoagulation (PRP) [Number; unit: Eyes] | 9

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Macular Edema
Description: Reduction in macular edema measured as
  * Proportion of eyes with baseline SD OCT CST >350 um demonstrating >15% reduction at week 52 from baseline
  * Proportion of eyes that demonstrate SD OCT CST <305um (males) and <290 um (females) at week 52 from baseline
Time Frame: 52 weeks from baseline
Population: Answered to the query of PRS review
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label Single Arm Trial
Number analyzed (Participants) | 30
Participants
  OCT CST >350 um demonstrating >15% reduction | 15
  OCT CST <305um (males): number analyzed (Participants) | 17
  OCT CST <305um (males) | 8
  OCT CST<290 um (females): number analyzed (Participants) | 13
  OCT CST<290 um (females) | 4

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Phase 4 Prospective, Nonrandomized, Open Label, Interventional
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 5/30
Other Adverse Events (participants affected / at risk) | 26/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 4 Prospective, Nonrandomized, Open Label, Interventional (N=30)
Hospitalization- Low electrolytes (Metabolism and nutrition disorders) | 1 (1)
Death (Cardiac disorders) | 1 (1) — Heart attack
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) — Hospitalized for sepsis
Kidney Failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 4 Prospective, Nonrandomized, Open Label, Interventional (N=30)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Common Cold (Infections and infestations) | 9 (9) — Including Influenzas, sinus infections, upper respiratory infections
Cardiovascular events (Cardiac disorders) | 1 (1) — Hypertension
Bladder Infection (Infections and infestations) | 1 (1)
Hernia (Gastrointestinal disorders) | 3 (3)
Blepharitis (Infections and infestations) | 1 (1)
Subconjunctival Hemorrhage (Eye disorders) | 2 (2)
Cataract Extraction (Surgical and medical procedures) | 1 (1)
Yag Laser Capsulotomy (Surgical and medical procedures) | 1 (1)
Trace Epiretinal Membrane (Eye disorders) | 1 (1)
Blurry Vision (Eye disorders) | 1 (1)
Kidney/Liver Conditions (Renal and urinary disorders) | 6 (6) — Kidney stone, bladder infection
Neurotoxicity (Nervous system disorders) | 1 (1)
Volume Overload (Renal and urinary disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size, no control group with continuation of bevacizumab/ranibizumab, 6 mth time point potentially skewed as last IAI at 4 mth due to protocol amendment. Loss of OCT, Fundus, Fluorescein Angiography on 1st 5 pts due to technical error

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/10/NCT03340610/Prot_SAP_000.pdf